CLINICAL TRIAL: NCT00492401
Title: Phase II Study of Decitabine in Acute Myeloid Leukemia
Brief Title: Decitabine in Treating Patients With Previously Untreated Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00246; OSU 07017; N01CM62207 (NIH)
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-05

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities | interventions — Decitabine; Chromatography, High Pressure Liquid; Microarray Analysis; Gene Expression Profiling; Mass Spectrometry; DNA Methylation

ARMS (1):
- Treatment (chemotherapy) (Experimental): Patients receive decitabine IV over 1 hour on days 1-10. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: decitabine; Other: laboratory biomarker analysis; Other: pharmacological study; Other: high performance liquid chromatography; Genetic: microarray analysis; Genetic: RNA analysis; Other: mass spectrometry; Genetic: DNA methylation analysis; Other: matrix-assisted laser desorption/ionization time of flight mass spectrometry

INTERVENTIONS:
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: high performance liquid chromatography — Correlative studies
  Other Names: HPLC
Genetic: microarray analysis — Correlative studies
  Other Names: gene expression profiling
Genetic: RNA analysis — Correlative studies
Other: mass spectrometry — Correlative studies
Genetic: DNA methylation analysis — Correlative studies
Other: matrix-assisted laser desorption/ionization time of flight mass spectrometry — Correlative studies
  Other Names: MALDI-TOF Mass Spectrometry

SUMMARY:
This phase II trial is studying how well decitabine works in treating patients with previously untreated acute myeloid leukemia. Drugs used in chemotherapy, such as decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the rate of complete remission (CR) in patients with previously untreated acute myeloid leukemia treated with decitabine.

SECONDARY OBJECTIVES:

I. Determine the rate of overall survival at 1 year in patients treated with this drug.

II. Determine the overall response rate (CR, incomplete CR, and partial remission) in patients treated with this drug.

III. Correlate the biological activity of decitabine with clinical endpoints and maximum concentration of plasma decitabine.

IV. Correlate intracellular concentration of decitabine with global DNA methylation, other biological endpoints, and clinical response.

OUTLINE:

Patients receive decitabine IV over 1 hour on days 1-10. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo bone marrow aspiration and blood sample collection periodically for pharmacological and correlative studies. Samples are analyzed for gene expression, methylation of gene promoters, fetal hemoglobin (HgF), DNMT1 protein expression, maximum concentration of plasma decitabine, and global DNA methylation. Samples are analyzed by RT-PCR, Bio-COBRA, matrix-assisted laser desorption ionization time-of-flight mass spectrometry, SDS-PAGE (polyacrylamide gel electrophoresis), immunoblotting, and LC-MS/MS.

After completion of study treatment, patients are followed for at least 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed acute myeloid leukemia (AML) meeting 1 of the following criteria:

  * At least 60 years of age and not a candidate for or refused standard induction treatment
  * Poor risk cytogenetics
  * AML following antecedent hematologic disorder
  * Therapy-related AML
  * Secondary AML
* No granulocytic sarcoma as sole site of disease
* No active CNS disease or CNS relapse
* ECOG performance status 0-2
* Life expectancy > 6 months
* Total bilirubin < 2.0 mg/dL
* Creatinine < 2.0 mg/dL
* AST and ALT < 2.5 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No NYHA class III or IV congestive heart failure
* No uncontrolled infection
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to decitabine that are not easily managed
* No other uncontrolled illness including, but not limited to, any of the following:

  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Serious cardiac arrhythmia
  * Psychiatric illness or social situations that would preclude compliance with study requirements
* No active second malignancy involving the blood or marrow or likely to progress and require therapy in the next 6 months
* No prior therapy for AML except emergency leukapheresis or hydroxyurea for leukocytosis
* No prior azacitidine or decitabine
* No prior cytarabine or other conventional chemotherapy agents for antecedent hematologic disorders

  * Prior myeloid growth factors, recombinant erythropoietin, thalidomide, or lenalidomide allowed
* No concurrent palliative radiotherapy
* No other concurrent investigational agents
* No other concurrent direct anti-leukemia therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-05; Primary Completion 2010-12 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Blum, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Blum W, Garzon R, Klisovic RB, Schwind S, Walker A, Geyer S, Liu S, Havelange V, Becker H, Schaaf L, Mickle J, Devine H, Kefauver C, Devine SM, Chan KK, Heerema NA, Bloomfield CD, Grever MR, Byrd JC, Villalona-Calero M, Croce CM, Marcucci G. Clinical response and miR-29b predictive significance in older AML patients treated with a 10-day schedule of decitabine. Proc Natl Acad Sci U S A. 2010 Apr 20;107(16):7473-8. doi: 10.1073/pnas.1002650107. Epub 2010 Apr 5. PMID 20368434

RESULTS

PARTICIPANT FLOW:
Groups:
- Decitabine: Decitabine 20mg/m2/day IV over 1 hour, days 1-10, repeat cycle every 28 days
Period: Overall Study
Arm/Group | Decitabine
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Decitabine
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 55
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: patients]
  United States | 54
  Canada | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Remission
Description: Per International Working Group criteria: Morphologic complete remission (CRm): Defined as morphologic leukemia-free state, including <5% blasts in BM aspirate with marrow spicules and a count of > 200 nucleated cells and no blasts with Auer rods, no persistent extramedullary disease, ANC > 1000/uL, platelet count > 100,000/uL. Patient must be independent of transfusions for a minimum of 1 week before each marrow assessment. Morphologic complete remission with incomplete blood count recovery (CRi): Defined as CR with the exception of neutropenia <1000/uL or thrombocytopenia <100,000/ul. Complete Remission Rate (CRm + CRi)
Time Frame: Up to 24 weeks
Measure: Number; unit: patients
Arm/Group | Decitabine
Number analyzed (Participants) | 55
patients | 25

2. Secondary Outcome: Measurement of DNA Methylation in Peripheral Blood or Bone Marrow Cells
Description: Standard paired statistical tests, parametric and nonparametric, will be used to baseline with treatment values. With data collected serially over time, repeated measures analysis of variance will be used to analyze data.
Time Frame: From baseline to up to day 28 of course 1
Population: Data was not collected and analyzed
Arm/Group | Decitabine
Number analyzed (Participants) | 0

3. Secondary Outcome: Measurement of DNMT Protein in Peripheral Blood or Bone Marrow Cells
Description: Expression studies were conducted using quantitative RT PCR. Expression of DNMT were normalized to the internal control to the ABL and levels of miR-29 to RNA U44.
Time Frame: Pre treatment
Population: Only pre treatment samples available for testing for 23 patients
Measure: Median (Inter-Quartile Range); unit: delta delta CT values
Groups:
- Responders: Any patient that achieved a CR (Complete Response), or Incomplete CR was categorized as a responder.
- Non Responder: Any patient that did not achieve a CR (Complete Response), or Incomplete CR was categorized as a non responder.
Arm/Group | Responders | Non Responder
Number analyzed (Participants) | 14 | 9
delta delta CT values
  Expression levels of MiR-29b | 0.0056394 [0.0037495 to 0.0075544] | 0.0024305 [0.0014533 to 0.0042197]
  Expression levels of DNMT3a | 0.000196066 [0.000145407 to 0.000280477] | 0.000341819 [0.000289839 to 0.000361753]
Statistical Analysis 1: Comparison: Responders vs Non Responder; Expression levels of miR-29b in pre treatment marrow samples from responding or non responding patients were compared using Wilcoxon rank sum tests; Test type: Superiority or Other; p = .02, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Responders vs Non Responder; Expression levels of DNMT3a in pre treatment marrow samples from responding or non responding patients were compared using Wilcoxon rank sum tests; Test type: Superiority or Other; p = .06, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Measurement of HbF in Peripheral Blood or Marrow Cells
Description: as for outcome 2
Time Frame: From baseline to up to days 28 of course 2
Population: Data was not collected and analyzed for this trial
Arm/Group | Decitabine
Number analyzed (Participants) | 0

5. Secondary Outcome: Measurement of Gene Expression in Peripheral Blood or Bone Marrow
Description: as for outcome 2
Time Frame: From baseline to up to day 28 of course 1
Population: Data was not collected and analyzed for this trial
Arm/Group | Decitabine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse events were graded according to the National Cancer Institute Common Toxicity Criteria for Adverse Events, version 3.0
Arm/Group | Treatment (Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 53/53
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy) (N=53)
Documented infection (Infections and infestations) | 31 (31) — Grade ≥ 3 in cycles 1 and 2
Febrile neutropenia (Infections and infestations) | 5 (5) — Grade ≥ 3 in cycles 1 and 2
Fatigue (General disorders) | 3 (3) — Grade ≥ 3 in cycles 1 and 2
Fever (General disorders) | 2 (2) — Grade ≥ 3 in cycles 1 and 2
Anorexia (Metabolism and nutrition disorders) | 1 (1) — Grade ≥ 3 in cycles 1 and 2
Dysgeusia (Nervous system disorders) | 1 (1) — Grade ≥ 3 in cycles 1 and 2
Mucositis/gingivitis (Gastrointestinal disorders) | 3 (3) — Grade ≥ 3 in cycles 1 and 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Grade ≥ 3 in cycles 1 and 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 (8) — Grade ≥ 3 in cycles 1 and 2
Prolonged QTc (Investigations) | 2 (2) — Grade ≥ 3 in cycles 1 and 2
Decreased left ventricular ejection fraction (Cardiac disorders) | 1 (1) — Grade ≥ 3 in cycles 1 and 2
Arrhythmia (Gastrointestinal disorders) | 3 (3) — Grade ≥ 3 in cycles 1 and 2
Hypertension (Vascular disorders) | 2 (2) — Grade ≥ 3 in cycles 1 and 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) — Grade ≥ 3 in cycles 1 and 2
Rash (Skin and subcutaneous tissue disorders) | 2 (2) — Grade ≥ 3 in cycles 1 and 2
Confusion (Psychiatric disorders) | 1 (1) — Grade ≥ 3 in cycles 1 and 2
Syncope (Nervous system disorders) | 3 (3) — Grade ≥ 3 in cycles 1 and 2
Abnormal gait (General disorders) | 2 (2) — Grade ≥ 3 in cycles 1 and 2
Pain (General disorders) | 7 (7) — Grade ≥ 3 in cycles 1 and 2
Thrombosis (Vascular disorders) | 3 (3) — Grade ≥ 3 in cycles 1 and 2
Hemorrhage/hematoma (Vascular disorders) | 5 (5) — Grade ≥ 3 in cycles 1 and 2

LIMITATIONS AND CAVEATS:
After completing the target accrual of 33 subjects, the study was expanded to include 22 additional patients. All patients who received decitabine are included in the analyses, except for two who had not completed therapy at the time of the analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days